CLINICAL TRIAL: NCT05757089
Title: An Open-label, Randomized, Cross-over, Comparative Study of ALCOFILTRUM Dietary Food Supplement for Alleviating Alcohol Hangover Symptoms in Healthy Volunteers
Brief Title: Efficacy of the Dietary Food Supplement ALCOFILTRUM in Alleviating Alcohol Hangover Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AVVA Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ALCOFILTRUM-NIR-B-07/2021
Record Dates: First submitted 2023-01-12; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Alcohol Drinking; Alcohol Intoxication
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALCOFILTRUM (Experimental): ALCOFILTRUM, 4 tablets in a single dose, 30 minutes prior to consumption of alcohol.
  Ingredients per tablet:
  Lignin hydrolyzed 800 mg; Glycine 150 mg; Dihydromyricetin 30 mg; Vitamin B1 30 mg.
  Interventions: Dietary Supplement: ALCOFILTRUM
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: ALCOFILTRUM — ALCOFILTRUM helps alleviate alcohol hangover symptoms after a single intake for 30 minutes before alcohol consumption.
  Arms: ALCOFILTRUM

SUMMARY:
The aim of this open-label, randomized, crossover, comparative pilot study is to assess efficacy and safety of the dietary food supplement ALCOFILTRUM in healthy volunteers who consume alcohol. Specifically the study will evaluate:

* Efficacy of the intervention to alleviate hangover symptoms in participants who consumed alcohol,
* Safety of intervention in participants who consuming alcohol.

Participants will take four tablets of ALCOFILTRUM dietary food supplement 30 minutes before alcohol ingestion, while the control group will intake only alcohol drink.

DETAILED DESCRIPTION:
Heavy drinking of alcoholic beverages may lead to hangover, characterized by a combination of unpleasant physical and mental symptoms that affect mood, cognition, and physical functioning. Hangover symptoms begin within several hours following drinking cessation, when a person's blood alcohol concentration (BAC) is falling, and peak when BAC is zero. The symptoms may continue for up to 24 hours thereafter. Multiple contributing factors are responsible for the development of alcohol hangover symptoms which include ethanol itself, its metabolites and congeners / fusel alcohols. The liver plays a key role in alcohol detoxification, and is therefore affected the most. Drinking large amounts of alcohol can lead to significant damage to the liver and brain cells, the reason for the need for protection.

In this open-label, randomized, cross-over, comparative pilot study investigators aim to assess efficacy and safety of the dietary food supplement ALCOFILTRUM in healthy volunteers who consume alcohol. Participants will consume an alcoholic drink (Bulbash Nano Original vodka 40%) in a dose calculated for every study subject based on ethanol 1.7g/kg body weight. The test group will take 4 tablets of ALCOFILTRUM dietary food supplement, 30 minutes before alcohol ingestion, while the control group will intake only alcohol drink. Twelve to thirteen hours after the last alcohol intake hangover symptoms will be evaluated based on questionnaires, and measurements of balance / coordination, attention and blood parameters. The findings from this study will provide important insight of a possible intervention for alleviating alcohol hangover symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged from 25 to 45 years inclusive.
* Body weight index of 18.5 to 30 kg/m2, with body weight of 60 kg to 100 kg.
* Healthy volunteers should behave adequately, with coherent speech observed.
* Available written Informed Consent for participation in this Study given by a healthy volunteer according to the effective laws.
* Subjects with history of episodic intake of alcohol and episodic hangover symptoms.
* Verified diagnosis "healthy": no chronic diseases in the history, no abnormal findings of lab tests and clinical investigations.

Exclusion Criteria:

* The Investigator's decision that a healthy volunteer is to be excluded in the interests of the volunteer.
* Any serious adverse event occurring to a healthy volunteer and associated with intake of alcohol and/or the study product.
* A healthy volunteer refusing to collaborate with the Medical Investigator or not complying with the Study procedure.
* A healthy volunteer was enrolled into the Study with violation of the Clinical Study Protocol.
* Any adverse events occurring to a healthy volunteer that, in a Medical Investigator's opinion, may endanger safety of a volunteer.
* Positive urine opioid test.
* Positive COVID-19 Ag Rapid Test.
* Positive blood alcohol test judging by concentration of alcohol fumes in exhaled air.
* 0.15 mg/L or higher content of alcohol fumes in exhaled air at the Screening Visit and at Visits 2, 3 prior to intake the first alcohol portion.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
1-item overall hangover severity rating | 13 hours
  Intensity of hangover symptoms in 12-13 hours after alcohol intake according to 1-item overall hangover severity rating. Score range is from 0 to 10, where higher scores mean more severe hangover symptoms.

SECONDARY OUTCOMES:
Schulte test | 13 hours
  Attention focusing and work efficiency according to Schulte test. Measurement timepoints: baseline, 1, 4, 12, 13 hours.
Romberg Stance test | 13 hours
  Coordination and stability assessment in Romberg Stances. Measurement coordination and stability timepoints: baseline, 1, 4, 12, 13 hours.
Mini Cog test | 13 hours
  Psychoneurological status. Measurement timepoints: baseline, 1, 4, 12, 13 hours.
Hangover Symptoms Questionnaire | 13 hours
  Score of Hangover Symptoms Questionnaire and frequency of hangover symptoms. Score rating from 0 to 4 for 24 diferent symptoms, where higher scores mean higher severity of the symptoms. Measurement timepoints: baseline, 1, 4, 12, 13 hours.
Blood Alcohol level | 12 hours
  Concentration of ethanol in per mille. Measurement timepoints: baseline, 1, 4, 12 hours.
Blood acetaldehyde level | 12 hours
  Concentration of acetaldehyde in ng/mL. Measurement timepoints: baseline, 1, 4, 12 hours.
C-reactive protein level | 12 hours
  Blood concentration of C-reactive protein in mg/L. Measurement timepoints: baseline, 4, 12 hours.
Bilirubin level | 12 hours
  Blood concentrations of bilirubin and bilirubin fractions (direct and indirect) in umol/L. Measurement timepoints: baseline, 12 hours.
Blood Inflamatory markers | 12 hours
  Concentrations of TNF-alpha and 8-isoprostane in pg/mL. Measurement timepoints: baseline, 4, 12 hours.
Liver enzyme markers | 12 hours
  Blood concentrations of AST, ALT, ALP, GGT in u/L. Measurement timepoints: baseline, 12 hours.

OTHER OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | 5 days
  Incidence rate of any adverse events.
Incidence of Serious Adverse events [Safety and Tolerability] | 5 days
  Incidence rate of any serious adverse events.
Arterial blood pressure [Safety and Tolerability] | 13 hours
  Level of systolic and diastolic arterial blood pressure 1; 2; 3, 4, 12, 13 hours vs. baseline.
Heart rate [Safety and Tolerability] | 13 hours
  Hear rate 1; 2; 3, 4, 12, 13 hours vs. baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Olga A. Sharapova, Ph.D., Principal Investigator — City Clinical Emergency Hospital
Locations (1):
- Clinical Emergency Hospital, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No